CLINICAL TRIAL: NCT02979587
Title: The Medtronic Harmony™ Transcatheter Pulmonary Valve Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Heart Valves (Industry)
Responsible Party: Sponsor
Organization: Medtronic Cardiovascular (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDT16004CON001
Record Dates: First submitted 2016-11-23; First posted 2016-12-01 (Estimated); Results first posted 2021-12-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Congenital Heart Disease; Tetrology of Fallot; RVOT Anomaly; Pulmonary Regurgitation
MeSH Terms: conditions — Heart Defects, Congenital; Tetralogy of Fallot; Pulmonary Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Harmony TPV System (Other): Intervention Device: Harmony Transcatheter Pulmonary Valves and Delivery Systems
  Interventions: Device: Harmony TPV System

INTERVENTIONS:
Device: Harmony TPV System — The Harmony™ TPV (Model NTPV0022) is comprised of a 22mm porcine pericardium valve, sewn to a polyester-covered nitinol frame.
  The Harmony TPV 25 and mTPV 25 (Model HTPV254952 and HTPV254252, respectively) is comprised of a 25mm porcine pericardium valve, sewn to a polyester covered asymmetrical hourglass nitinol frame with larger diameter inflow and outflow as well as shorter length compared to TPV 22 (Harmony TPV 25 Model HTPV254952 is not applicable for Continued Clinical Experience).
  The Harmony Delivery System (DS) for the TPV 22, TPV 25, and mTPV 25 (NTPVDS0022 and HTPVDS0025) are all 25 Fr delivery systems using a coil loading catheter.

SUMMARY:
The purpose of this study is to further evaluate the safety and effectiveness of the Harmony™ TPV system. The Pivotal/CAS phases of the study have transitioned into a post-approval study to confirm the long-term functionality of transcatheter implantation of the Medtronic Harmony TPV.

DETAILED DESCRIPTION:
The continued clinical experience addendum is a prospective, multi-center, non-randomized, interventional study to evaluate the safety and effectiveness of the Harmony TPV system. All implanted subjects will receive the Harmony TPV 22 or Harmony mTPV 25 device. This phase allows up to 45 subjects implanted with TPV 22 in the United States and Canada, and up to 84 subjects implanted with mTPV 25 in the United States.

The Post Approval Phase (PAS) addendum is a prospective, multi-center, non-randomized, post-market study to evaluate the safety and effectiveness of the Harmony TPV system in the United States. All implanted subjects have been implanted with the Harmony TPV 22 or Harmony mTPV 25 device during the pivotal or CAS phase of the study. The PAS addendum extends follow-up from five years to ten years for consenting subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has severe pulmonary regurgitation as assessed via echocardiography or CMR determined PR fraction >/= 30%
* Subject has clinical indication for surgical placement of an RV-PA conduit or bioprosthetic pulmonary valve
* Subject is willing to consent to participate

Exclusion Criteria:

* Patients with right ventricular outflow tract obstruction (RVOTO) lesions surgically treated with an RV-to-PA conduit implant
* RVOT anatomy or morphology that is unfavorable for device anchoring
* Positive pregnancy test
* Life expectancy of less than 1 year

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2031-02 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John P Cheatham, MD, Principal Investigator — Nationwide Children's Hospital
Locations (12):
- United States (9):
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Mayo Clinic, Rochester, Minnesota
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Canada (2):
  - The Hospital for Sick Children (SickKids), Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
- National Cerebral and Cardiovascular Center, Suita, Osaka, Japan

REFERENCES:
- [Derived] Morray BH, Gillespie MJ, Cheatham JP, Salavitabar A, Peng L, Jones TK, Levi DS, Gray RG, Asnes J, Cabalka AK, Fujimoto K, Qureshi AM, Bergersen L, Benson LN, Haugan D, McElhinney DB. Midterm Outcomes in a Pooled Cohort of Harmony Transcatheter Pulmonary Valve Recipients. Circ Cardiovasc Interv. 2025 Sep;18(9):e015196. doi: 10.1161/CIRCINTERVENTIONS.125.015196. Epub 2025 Jul 16. PMID 40665900
- [Derived] Gillespie MJ, Bergersen L, Benson LN, Weng S, Cheatham JP. 5-Year Outcomes From the Harmony Native Outflow Tract Early Feasibility Study. JACC Cardiovasc Interv. 2021 Apr 12;14(7):816-817. doi: 10.1016/j.jcin.2021.01.046. No abstract available. PMID 33826508

RESULTS

PARTICIPANT FLOW:
Groups:
- Implanted Pivotal Harmony TPV Subjects: This study is comprised of a single arm of subjects implanted with the Harmony TPV device during the pivotal study.
Period: Overall Study
Arm/Group | Implanted Pivotal Harmony TPV Subjects
Started (Number of subject implanted) | 50
Catheterized (Number of subjects catheterized with the intent to implant Harmony TPV) | 50
Implanted (Number of subjects implanted with a Harmony TPV) | 50
Implanted > 24 Hours (Number of subjects implanted successfully for at least 24 hours) | 48
Completed (Subjects with evaluable data at 6 months) | 48
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Harmony Pivotal Subjects- Catheterized Cohort
Arm/Group | Implanted Pivotal Harmony TPV Subjects
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 40
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 48
  Japan | 2

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Procedure- or Device-related Mortality at 30 Days.
Description: The primary safety endpoint is point estimate of freedom from procedure or device-related mortality rate at 30 days post procedure.
Time Frame: 30 days
Population: The catheterized cohort consists of all subjects who undergo catheterization for possible implantation of the Harmony TPV. The primary safety endpoint population includes all subjects that were catheterized and also had evaluable data at 30 days. Two subjects were exited prior to the 30 day timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Catheterized Cohort: Subjects included in this analysis were those who were catheterized for a Harmony TPV implant and had evaluable data at 30 days.
Arm/Group | Catheterized Cohort
Number analyzed (Participants) | 48
Participants | 48

2. Primary Outcome: Number of Participants With Acceptable Hemodynamic Function Composite at 6 Months
Description: Defined as:
  * Mean RVOT gradient as measured by continuous-wave Doppler ≤40 mmHg -AND-
  * Pulmonary regurgitant fraction as measured by magnetic resonance imaging <20%
Time Frame: 6 months
Population: The implanted >24 hours cohort consists of all subjects who have a Harmony TPV implanted which remains implanted for greater than 24 hours.
Measure: Count of Participants; unit: Participants
Groups:
- Implanted > 24 Hours Cohort: Subjects included in this analysis were those who were successfully implanted with a Harmony TPV for greater than 24 hours and had evaluable data at 6 months.
Arm/Group | Implanted > 24 Hours Cohort
Number analyzed (Participants) | 48
Participants | 43

3. Secondary Outcome: Number of Participants With Technical Success at Exit From Catheterization Lab/Operating Room (OR)
Description: Technical success at exit from catheterization lab/operating room (OR), as defined as:
  * No device- or procedural-related mortality, with
  * Successful access, delivery and retrieval of the delivery system, and
  * Deployment and correct positioning (including minor repositioning if needed) of the single intended device, and
  * No need for additional unplanned or emergency surgery or re-intervention related to the device or access procedure
Time Frame: At exit from catheterization lab/operating room (OR)
Population: The attempted implant cohort consists of all subjects who undergo catheterization and a Harmony TPV implantation was attempted (Harmony TPV is introduced into the subject's body).
Measure: Count of Participants; unit: Participants
Groups:
- Attempted Implant Cohort: Subjects included in this analysis were those who had an attempted Harmony TPV implant
Arm/Group | Attempted Implant Cohort
Number analyzed (Participants) | 50
Participants | 45

4. Secondary Outcome: Device Success Out to 5 Years
Description: Device success is defined as:
  * No device- or procedural-related mortality, with
  * Original intended device in place, and
  * No additional surgical or interventional procedures related to access or the device since completion of the original procedure (i.e., exit from the catheterization lab), and
  * Intended performance of the device, as defined as:
    * Structural performance: No migration, embolization, detachment, major stent fracture, hemolysis, thrombosis, endocarditis, and
    * Hemodynamic performance: Relief of insufficiency (PR < moderate) without producing the opposite (mean RVOT gradient > 40 mmHg) as measured by continuous wave Doppler, and
  * Absence of para-device complications, as defined by:
    * PVL = moderate, or
    * Erosion, or
    * RVOT or PA rupture
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2026-04

5. Secondary Outcome: Number of Participants With Procedural Success at 30 Days
Description: Procedural success is defined as:
  * Device success at 30 days, and
  * None of the following device- or procedure-related serious adverse events:
    * Life-threatening major bleed
    * Major vascular or cardiac structural complications required unplanned reintervention or surgery
    * Stage 2 or 3 acute kidney injury (AKI) (includes new dialysis)
    * Pulmonary embolism
    * Severe heart failure (HF) or hypotension requiring IV inotrope, ultrafiltration, or mechanical circulatory support
    * Prolonged intubation >48 hours
Time Frame: 30 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Attempted Implant Cohort
Number analyzed (Participants) | 50
Participants | 42

6. Secondary Outcome: Freedom From TPV Dysfunction Out to 5 Years
Description: TPV dysfunction is defined as any one of the following:
  * RVOT reoperation for device-related reasons
  * Catheter re-intervention of TPV
  * Hemodynamic dysfunction of the TPV (moderate or greater pulmonary regurgitation, and/or a mean RVOT gradient >40 mmHg)
Time Frame: 5 years (5 year data has an anticipated reporting date of April 2026)
Reporting Status: Not Posted, anticipated posting 2026-04

7. Secondary Outcome: Assessment of Safety
Description: All procedure-related serious adverse events. All device-related serious adverse events. Death (all-cause, procedural, and device-related).
Time Frame: Ongoing
Reporting Status: Not Posted

8. Secondary Outcome: Characterization of Quality of Life Scores Out to 5 Years
Description: Quality of life score over time will be assessed by the SF-36 at pre-implant, 1 month post-implant, 6 months post-implant, 1 year post-implant, 2 years post-implant, and 3 years. The analysis cohort will be the implanted > 24 hours cohort. Minimum score of 0 and maximum score of 100 is possible. Higher values are considered to be a better outcome.
Time Frame: Baseline, 30 Day, 6 Month, 1 Year, 2 Year, 3 Year
Population: Number analyzed differs from overall number analyzed because subjects have either exited or have not yet completed that timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Implanted > 24 Hours Cohort: Subjects included in this analysis were those who were successfully implanted with a Harmony TPV for greater than 24 hours and had evaluable data at the given timepoint.
Arm/Group | Implanted > 24 Hours Cohort
Number analyzed (Participants) | 48
score on a scale
  Baseline | 80.5 (25.6)
  30 Day Follow-up: number analyzed (Participants) | 46
  30 Day Follow-up | 90.2 (15.6)
  6 Month Follow-up: number analyzed (Participants) | 45
  6 Month Follow-up | 94.6 (8.8)
  1 Year Follow-up: number analyzed (Participants) | 44
  1 Year Follow-up | 91.6 (14.9)
  2 Year Follow-up: number analyzed (Participants) | 24
  2 Year Follow-up | 94.4 (11.0)
  3 Year Follow-up: number analyzed (Participants) | 6
  3 Year Follow-up | 98.3 (4.1)

9. Secondary Outcome: Characterization of Right Ventricle Remodeling Following TPV Implant
Description: Right ventricle remodeling will be assessed via CMR at pre-implant and 6 months post-implant. The analysis cohort will be implanted longer than 24 hours cohort. The characterization will be made using right ventricular end diastolic volume (ml).
Time Frame: Baseline, 6 Month
Population: Subjects included in this analysis were those who were successfully implanted with a Harmony TPV for greater than 24 hours and had evaluable CMR data at the given timepoint.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Implanted > 24 Hours Cohort
Number analyzed (Participants) | 26
ml
  Pre-implant | 291.5 (57.4)
  6 Months | 223.0 (54.9)

10. Secondary Outcome: Characterization of Quality of Life Scores Out to 5 Years
Description: Quality of life score over time will be assessed by the SF-36 at 4 & 5 years. The analysis cohort will be the implanted > 24 hours cohort. Minimum score of 0 and maximum score of 100 is possible. Higher values are considered to be a better outcome.
Time Frame: 4 Year, 5 Year (4 & 5 year data has an anticipated reporting date of April 2026)
Reporting Status: Not Posted, anticipated posting 2026-04

11. Secondary Outcome: Characterization of Right Ventricle Remodeling Following TPV Implant
Description: Right ventricle remodeling will be assessed via CMR at 2 years post- implant and 5 years post-implant. The analysis cohort will be implanted longer than 24 hours cohort. The characterization will be made using right ventricular end diastolic volume (ml).
Time Frame: 2 Year, 5 Year (2 & 5 year data has an anticipated reporting date of April 2026)
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: Adverse Event data are collected through study completion, an average of 5 years
Description: Serious Adverse Event:
  1. led to death,
  2. led to a serious deterioration in the health of the subject, resulting in
     1. a life-threatening illness or injury or
     2. a permanent impairment of a body structure or a body function or
     3. in-patient or prolonged hospitalization or
     4. medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function
  3. led to foetal distress, death or congenital abnormality/birth defect.
Groups:
- Catheterized Cohort: The catheterized cohort consists of all subjects who undergo catheterization for possible implantation of the Harmony TPV.
Arm/Group | Catheterized Cohort
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 3/50
Other Adverse Events (participants affected / at risk) | 33/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheterized Cohort (N=50)
Complete Heart Block (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (Cardiac disorders) | 1 (1)
Device Dislocation (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Catheterized Cohort (N=50)
Arrhythmia (Cardiac disorders) | 4 (4)
Palpitations (Cardiac disorders) | 3 (3)
Premature Ventricular Ectopic Beats (Cardiac disorders) | 6 (6)
Supraventricular Tachycardia (Cardiac disorders) | 3 (3)
Tricuspid Regurgitation (Cardiac disorders) | 3 (3)
Ventricular Tachycardia (Cardiac disorders) | 7 (7)
Vomiting (Gastrointestinal disorders) | 3 (3)
Chest Pain (General disorders) | 6 (6)
Fever (General disorders) | 10 (13)
Radiation Burn (Injury, poisoning and procedural complications) | 3 (4)
Device Shape Alteration (Product Issues) | 3 (3)
Paravalvular Leak (Product Issues) | 5 (5)
Hemorrhage (Vascular disorders) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/87/NCT02979587/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT02979587/SAP_002.pdf